CLINICAL TRIAL: NCT03984565
Title: PAIN: a Project Assessing the Impact of a Novel Cannabinoid Product
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Staci Gruber, Ph.D. (Other)
Collaborators: Etheridge Foundation (Unknown)
Responsible Party: Sponsor-Investigator, Staci Gruber, Ph.D., Director, Marijuana Investigations for Neuroscientific Discovery; Director, Cognitive and Clinical Neuroimaging Core; Associate Professor of Psychiatry, Harvard Medical School, Mclean Hospital
Organization: Mclean Hospital (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2023P001774
Record Dates: First submitted 2019-06-07; First posted 2019-06-13 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Chronic Pain
Keywords: Cannabidiol; Medical Cannabis; Industrial Hemp
MeSH Terms: conditions — Chronic Pain | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cannabidiol Treatment Arm (Experimental): High-CBD sublingual product administered three times daily for the treatment period.
  Interventions: Drug: Cannabidiol
- Placebo Treatment Arm (Placebo Comparator): Placebo sublingual product administered three times daily for the treatment period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cannabidiol — High-CBD, low-THC sublingual product formulated in palm oil
  Other Names: CBD
  Arms: Cannabidiol Treatment Arm
Drug: Placebo — Placebo sublingual product formulated in palm oil with supplemental terpenes to match CBD product.
  Arms: Placebo Treatment Arm

SUMMARY:
This study is a clinical trial of a high-cannabidiol (CBD) sublingual product compared to placebo for 9 weeks in patients with chronic pain conditions. The study will assess the impact of CBD on chronic pain symptoms, conventional medication use, clinical state, quality of life, cognition, and biomarkers.

DETAILED DESCRIPTION:
Cannabis sativa has been used medicinally to treat a wide range of disorders for thousands of years. Cannabis is comprised of more than 100 cannabinoids, including D9-tetrahydrocannabinol (THC), the major intoxicating constituent, and cannabidiol (CBD), the major non-intoxicating constituent that has a number of potential therapeutic properties. Although a wide range of medical cannabis (MC) and hemp products (containing less than 0.3% THC) are used by consumers for a variety of medical indications, little is known about the direct impact of individual cannabinoids and constituent ratios on the symptoms that cause patients to seek treatment.

Chronic pain is one of the most common indications for MC use, and several studies have yielded compelling data suggesting that MC and its constituents may have analgesic and anti-inflammatory properties, suggesting that cannabinoids may have the potential to treat chronic pain. This investigation will involve a placebo-controlled crossover trial of a hemp-derived high-CBD, low-THC sublingual product in patients with chronic pain; patients will be assessed at baseline and over 69weeks of treatment with CBD or placebo on measures of clinical state, including pain and related symptoms, conventional medication use, and cognition, and provide samples for analysis of inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent
* Subject is 21 or older
* Subject is fluent in English
* Subject endorses a musculoskeletal chronic pain condition including, but not limited to, chronic pain due to injury, arthritis (including osteoarthritis and rheumatoid arthritis), bursitis, etc.

Exclusion Criteria:

* Non-fluent English speakers
* Estimated IQ < 75
* A history of head injury or loss of consciousness greater than 5 minutes
* Currently uses CBD products regularly
* Female subjects will be excluded if they have a positive urine pregnancy test, are trying to become pregnant, or are currently breastfeeding
* Presence of a serious or unstable medical illness, including liver, kidney, or cardiovascular disease (hyper/hypotension, cardiac disorders), or neurological disorder (including seizure disorder)
* Primary neuropathic pain or cancer-related pain; patients experiencing neuropathic pain secondary to musculoskeletal pain will be allowed to enter the study
* Disclosure of a genetic polymorphism affecting CYP2C9 function

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-06-27 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in pain ratings on a Numerical Rating Scale (NRS) | 6 weeks
  The NRS is an 11-point scale on which subjects rate their pain by choosing a number between 0 (no pain) and 10 (worst possible pain). Lower scores indicate less pain.

SECONDARY OUTCOMES:
Change in pain ratings on the Brief Pain Inventory (BPI) | 6 weeks
  The BPI contains 9 questions that assess the severity of pain, how much relief is provided by treatment, and the functional impact of the pain within the last 24 hours. Lower scores are better.
Change in ratings on the Pain Self-Efficacy Questionnaire (PSEQ) | 6 weeks
  The PSEQ contains several questions assessing the patients' confidence in carrying out certain activities despite their pain on a 7-point scale ranging from 0 (not at all confident) to 6 (completely confident). Higher scores are better.
Change in ratings on the Pain Distress Scale (PDS) | 6 weeks
  The PDS is an 11-point scale one where subjects rate their pain by level of distress the pain causes on a scale of 0 to 10. Lower scores are better.
Change in ratings on the Pain Disability Index (PDI) | 6 weeks
  On the PDI, the subject rates how their pain affects 7 different areas of their life on a scale of the level of disability that their pain causes, from "no disability" to "worst disability". Lower scores are better.
Change in Conventional Medication Use | 6 weeks
  Change in conventional medication use, including opioids, will be assessed and analyzed. Changes in dose and frequency of conventional medication use will be quantified.

CONTACTS AND LOCATIONS:
Overall Officials: Staci Gruber, Ph.D., Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided